CLINICAL TRIAL: NCT00692926
Title: A Pilot Trial of Unrelated Umbilical Cord Blood Transplantation Augmented With Ex Vivo CytokinePrimed ALDHbr Umbilical Cord Blood Cells
Brief Title: Unrelated Umbilical Cord Blood Transplantation Augmented With ALDHbr Umbilical Cord Blood Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joanne Kurtzberg, MD (Other)
Collaborators: Aldagen (Industry)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008970; 7177 (Other: Legacy IRB number)
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: MDS; Anemia, Aplastic; Inborn Errors of Metabolism; Congenital Marrow Failure; Congenital Immunodeficiency Syndrome
Keywords: ALDHbr; Umbilical Cord Blood; Transplantation; Hematological malignancy; MDS; severe aplastic anemia; inborn error of metabolism; congenital marrow failure or congenital immunodeficiency syndrome; Hurler's Disease; Tay Sach's; PMD; Hunter's Syndrome; Krabbe; MLD; ALD; ALL; AML
MeSH Terms: conditions — Anemia, Aplastic; Metabolism, Inborn Errors; Primary Immunodeficiency Diseases; Hematologic Neoplasms; Mucopolysaccharidosis I; Mucopolysaccharidosis II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 20% primed UCB (Other): 20% of UCB is ALDHbr sorted and primed and give on transplant day after conventional graft
  Interventions: Biological: ALDHbr Umbilical Cord Blood Cells
- 20% un-primed (Other): 20% of UCB is ALDHbr freshly sorted and give on transplant day 4-8 hrs after conventional graft
  Interventions: Biological: ALDHbr Umbilical Cord Blood Cells
- Double- 1 unit primed (Other): patient receives 1 conventional UCB unit and 1 unit that has been ALDHbr sorted and primed
  Interventions: Biological: ALDHbr Umbilical Cord Blood Cells
- Double- 1 unit unprimed (Other): Patient receives 1 UCB unit and a second UCB unit that has been freshly ALDHbr sorted
  Interventions: Biological: ALDHbr Umbilical Cord Blood Cells

INTERVENTIONS:
Biological: ALDHbr Umbilical Cord Blood Cells — ALDHbr sorted Umbilical Cord Blood Cells

SUMMARY:
The main purpose of this investigational (not approved by the FDA) Phase I research is to test whether transplantation of umbilical cord blood cells can be safely supplemented with a transfusion of a portion of these cells that have been sorted (collected from a special machine called a cell sorter) and then either infused a few hours after the standard transplant or for some patients grown in a special system in the laboratory prior to the transplant, designed to increase the number of stem cells transplanted. This system is currently in the early phases of testing.

DETAILED DESCRIPTION:
The main purpose of this study is to test whether transplantation of umbilical cord blood cells can be safely supplemented with transfusion of a portion of these cells that have been grown in a special system (designed to increase the number of cells transplanted) in the laboratory prior to the transplant. This system is currently in the early phases of testing in a FDA-IND-sponsored clinical trial. If the patient consents to participate in this study, approximately 1/5th (20%) of the cord blood unit selected for the transplant will be treated per protocol. The first 3 patients will receive ALDHbr sorted cells but not primed in culture. This is to test the safety of the ALDHbr cells. The treated cells will be given to the patient on the day of transplant approximately 4 hours after the standard or conventional transplant which will be given from the 80% fraction of the cord blood unit. A total of 26 evaluable patients are to be enrolled as outlined below (protocol has been amended to allow this enrollment):

* 10 evaluable patients who received ALDHbr freshly sorted cells (20% portion)
* 10 evaluable patients who received ALDHbr sorted and cytokine primed cells (20% portion)
* 3 evaluable patients who received a conventional cord blood unit and a cord blood unit that has been ALDHbr sorted (sort of the UCB unit will be done on Day -1 due to the time it takes to actually perform the sort)
* 3 evaluable patients who received a conventional cord blood unit and a cord blood unit that has been ALDHbr sorted and cytokine primed (sort and priming will be done on day -5 as described later in the protocol)

ELIGIBILITY:
Inclusion Criteria:

-Hematologic Malignancy: High risk ALL in first complete remission ALL or ANLL in second or subsequent remission ANLL in relapse MDS CML in any chronic phase or accelerated phase Severe aplastic anemia refractory to medical therapy The subject is negative for CNS disease at time of enrollment.

* Inborn errors of metabolism Hurler Syndrome (MPS I) Hurler-Scheie Syndrome Hunter Syndrome (MPS II) Sanfilippo Syndrome (MPS III) Morquio Syndrome (MPS IV) Maroteaux-Lamy Syndrome (MPS VI) Krabbe Disease (Globoid Leukodystrophy) Metachromatic Leukodystrophy (MLD) Adrenoleukodystrophy(ALD and AMN) Sandhoff Disease Tay Sachs Disease The subject does NOT have uncontrolled seizures, apnea, evidence of aspiration pneumonia or evidence of brain stem involvement on MRI scans
* Congenital marrow failure Amegakaryocytic thrombocytopenia TAR Kostmann's Syndrome Schwachman-Diamond Syndrome Blackfan-Diamond Anemia
* Congenital immunodeficiency syndromes requiring myeloablative therapy Wiscott Aldrich Syndrome LAD CGD FEL/HLH CVID/CID
* SUBJECT'S DONOR Subject does NOT have a 6/6 or 5/6 antigen matched related bone marrow donor. Suitably matched cord blood unit with adequate cell dose is available. Unit must be in a dual compartment bag.

PERFORMANCE STATUS and ORGAN FUNCTION

* <55 years of age at time of enrollment.
* Lansky score between 60% and 100%, or a Karnofsky score between 50% and 100%
* Adequate function of other organ systems
* Creatinine < 2.0 mg/dl and creatinine clearance > 50 cc/min/m2
* Hepatic transaminases (ALT/AST) < 4 x normal, bilirubin < 2.0 mg/dl
* Normal cardiac function by echocardiogram or radionuclide scan
* Pulmonary function tests demonstrating FVC, CVC, and FEV1 of >60% of predicted for age. For adult patients DLCO > 60% of predicted. If patient cannot perform PFTs, clearance by the pediatric or adult pulmonologist will be required
* No uncontrolled infections at the time of cytoreduction
* NOT pregnant or lactating (must have a current negative pregnancy test)
* HIV negative
* Subject is not concurrently involved in any other clinical trial that affects engraftment or immune reconstitution (e.g. other hematopoietic growth factors).
* Subject does not have any co-morbid condition, which in the view of the Principal Investigators, renders the patient at too high a risk from treatment complications and regimen related morbidity/mortality.

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2005-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To assess the safety of infusing ex vivo cytokine-primed ALDHbr cells isolated from banked unrelated umbilical cord blood (CB) into patients also receiving a standard unmanipulated unrelated CB transplant delivering >2.5x10e7 nucleated cells per kg. | Prospective

SECONDARY OUTCOMES:
To describe the biological effect of ex vivo cytokine-primed ALDHbr cells in these patients on neutrophil and platelet engraftment and immune reconstitution. | prospective
To describe the clinical outcomes in these patients: - incidence of infections -Non relapse mortality -incidence of acute and chronic graft-vs-host disease -overall survival at 180 days | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States